CLINICAL TRIAL: NCT03796403
Title: Comparison of Bupivacaine Peritoneal Infiltration and Intramuscular Diclofenac Versus Bupivacaine Peritoneal Infiltration Alone for Postoperative Pain Relief in Gynecologic Cancer Patients Undergoing Open Surgery
Brief Title: Bupivacaine Plus Diclofenac Versus Bupivacaine Alone for Postoperative Pain Relief in Gynecologic Cancer Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Diclofenac is no longer recommend for intramuscular administration by the Medical Council of Thailand
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Suphetgyn2516
Record Dates: First submitted 2018-09-28; First posted 2019-01-08 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2019-01

CONDITIONS: Post-operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Diclofenac

STUDY DESIGN:
Intervention Model Description: randomized into two groups by simple random. In bupivacaine and diclofenac group (n=70), Twenty ml of bupivacaine was infiltrated into surgical-site peritoneum and diclofenac 75 mg was intramuscularly injected immediately after complete the procedure and the operative field was covered with sterile adhesive wound dressing. In the bupivacaine alone group (n=70), 20 ml of bupivacaine was infiltrated into surgical-site peritoneum before closure and a 3 ml of sterile water was intramuscularly injected immediately after complete the procedure. Intravenous morphine injection was given if the pain score was more than 6 in the first 24 hours. Post-operation; time to first request of pain medication, doses, side effects, and vital signs were recorded. VAS was recorded at 2, 6, 12 and 24 hours post-operation and patients' satisfied score was recorded after 24 hours post-operation.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- diclofenac and bupivacaine group (Experimental): Twenty mL of bupivacaine was infiltrated into surgical-site peritoneum , divided in 10 sites before closure, and diclofenac 75 mg (3 mL) was intramuscularly injected immediately after complete the procedure and the operative field was covered with sterile adhesive wound dressing.
  Interventions: Other: Diclofenac
- bupivacaine only group (Placebo Comparator): Twenty mL of bupivacaine was infiltrated into surgical-site peritoneum, divided in 10 sites before closure and a 3 mL of sterile water was intramuscularly injected immediately after complete the procedure.
  Interventions: Other: Diclofenac

INTERVENTIONS:
Other: Diclofenac — Twenty mL of bupivacaine was infiltrated into surgical-site peritoneum , divided in 10 sites before closure, and diclofenac 75 mg (3 mL) was intramuscularly injected immediately after complete the procedure and the operative field was covered with sterile adhesive wound dressing.

SUMMARY:
compare the postoperative pain between Bupivacaine peritoneal Infiltration plus immediately postoperative intramuscular Diclofenac and Bupivacaine peritoneal infiltration alone by using visual analogue score (VAS).

DETAILED DESCRIPTION:
The primary objective is to compare the postoperative pain between Bupivacaine peritoneal Infiltration plus immediately postoperative intramuscular Diclofenac and Bupivacaine peritoneal infiltration alone by using visual analogue score (VAS). The secondary objective is to evaluate the time to first dose and the total amount of morphine requirement after the operation in both groups.

ELIGIBILITY:
Inclusion Criteria:

* gynecologic cancer patients ,i.e. cervical cancer, endometrial cancer, or ovarian tumor suspicious for malignancy
* who has scheduled for operation via laparotomy route
* Women who has ASA physical status I-II
* All of the have age more than 20 years old
* able to communicate in Thai
* Women who agrees to participate in this study

Exclusion Criteria:

* patient who had emergency conditions - indication for emergency operation
* intraoperative cardiac arrhythmia
* operation purpose for only tumor biopsy

  * Women who have abnormal kidney function test (Cr > 1.5)
  * Women with history of gastrointestinal bleeding
  * Women who take the antiplatelet or anticoagulant medications
  * Women with history of allergy to bupivacaine and NSAIDs
  * Women who cannot evaluated pain score

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Gynecologic cancer patients
Enrollment: 140 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Post-operative pain relief | During acute post operation peroid as 24 hours post operation
  compare the postoperative pain between Bupivacaine peritoneal Infiltration plus immediately postoperative intramuscular Diclofenac and Bupivacaine peritoneal infiltration alone by using visual analogue score(VAS). Score 0-10 .When Score is higher than 5 score ,the pateint will gain the analgesia as opioid.

SECONDARY OUTCOMES:
Morphine requirement | During acute post operation period as 24 hours post operation
  evaluate the time to first dose post operation and the total amount of morphine requirement after the operation in both groups. Score 0-10 .When Score is higher than 5 score ,the pateint will gain the analgesia as opioid.

CONTACTS AND LOCATIONS:
Overall Officials: Suphet Tuipae, MD, Principal Investigator — Department of Medical Services Ministry of Public Health of Thailand
Locations (1):
- Rajavithi hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No